CLINICAL TRIAL: NCT00682344
Title: Pharmacokinetic of levobupivacaïne After Sciatic Nerve Block in Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2007-000796-42; 2007-08
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Surgical Pathology of the Leg or the Foot.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levobupivacaïne — 1,75mg/kg

SUMMARY:
Levobupivacaïne (Chirocaine®) is a new local anaesthetic recently marketed in France. The goal of this prospective work is to study the pharmacokinetic aspect of this drug after injection around the sciatic nerve (subgluteal way).

DETAILED DESCRIPTION:
The originality of this work is to call upon a modelling of pharmacokinetic by using the principle of the pharmacology of population.

This work also proposes to appreciate a dynamic aspect since data of effectiveness and tolerance will be collected with regular intervals during the first 24 hours after the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Surgical pathology of the leg or the foot with garot tyre of thigh
* Age included between 6 months and 12 years
* Status ASA I or II

Exclusion Criteria:

* Bilateral or one-sided surgical gesture realized without garot tyre
* Cutaneous infection in the point of draining
* Clinical confusion of the coagulation
* Allergy informed in the local anesthesics of amino-acid class
* Evolutionary neurological pathology of the operated limb
* Renal, respiratory, cardiac or hepatic insufficiency.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The purpose of this work is to describe the pharmacokinetics characteristics by the levobupivacaine after peripheral block by using the principle of the pharmacology of population, this allowing fewer sampling of blood by patients. | 24 months

SECONDARY OUTCOMES:
Appreciation, by the anaesthetist in charge of the patient, of the quality of the "surgical" analgesia during the surgery by: very effective, effective, ineffective. Measure of the delay of appeal of the first one bolus of morphine. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric LACROIX, MD, Principal Investigator — ASSISTANCE PUBLIQUE DES HOPITAUX DE MARSEILLE
Locations (1):
- Hôpital de la Timone - Pôle d'anesthésie réanimation pédiatrique, Marseille, France